CLINICAL TRIAL: NCT06081322
Title: An Exploratory Study to Evaluate the Safety and Efficacy of Peptide Receptor Radionuclide Therapy With 177Lu-EB-FAPI in Patients With Advanced Cholopancreatic Tumors
Brief Title: A Study to Evaluate the Safety and Efficacy of PRRT With 177Lu-EB-FAPI in Patients With Advanced Cholopancreatic Tumors
Acronym: CISPD-5
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CISPD-5
Record Dates: First submitted 2023-06-12; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-06

CONDITIONS: Advanced Pancreatic Cancer and Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase Ia: Dose escalation (Experimental): To determine the therapeutic dose of 177Lu-EB-FAPI using a 3 + 3 dose-escalation mode
  Interventions: Drug: PRRT with 177Lu-EB-FAPI
- Phase Ib: Dose expansion-pancreatic cancer cohort (Experimental): In pancreatic cancer cohort, patients will receive the first phase determined dose of 177Lu-EB-FAPI every 4 weeks, and each patient will receive no more than 4 cycles.
  Interventions: Drug: PRRT with 177Lu-EB-FAPI
- Phase Ib: Dose expansion-cholangiocarcinoma cohort (Experimental): In cholangiocarcinoma cohort, patients will receive the first phase determined dose of 177Lu-EB-FAPI every 4 weeks, and each patient will receive no more than 4 cycles.
  Interventions: Drug: PRRT with 177Lu-EB-FAPI

INTERVENTIONS:
Drug: PRRT with 177Lu-EB-FAPI — PRRT with 177Lu-Fibroblast activation protein inhibitor and modified by Evans blue

SUMMARY:
This study is a prospective, single-center, open, single-arm, exploratory study to evaluate the safety and efficacy of 177Lu-EB-FAPI PRRT, and to explore 177Lu-EB-FAPI in patients with advanced pancreatic cancer and cholangiocarcinoma. Eligible patients with advanced pancreatic cancer or cholangiocarcinoma were screened and enrolled after signing the informed consent forms. In the first stage of the enrolled patients, the 177Lu-EB-FAPI treatment dose was determined using a 3 + 3 dose escalation mode. Patients enrolled in the second phase, divided into pancreatic cancer cohort and cholangiocarcinoma based on pathology, will receive the first phase determined dose of 177Lu-EB-FAPI every 4 weeks, and each patient will receive no more than 4 cycles. The aim of the study is to evaluate the safety and efficacy of the 177Lu-EB-FAPI treatment.

DETAILED DESCRIPTION:
This study is a prospective, single-center, open, single-arm, exploratory study to evaluate the safety and efficacy of 177Lu-EB-FAPI PRRT, and to explore 177Lu-EB-FAPI in patients with advanced pancreatic cancer and cholangiocarcinoma. Eligible patients with advanced pancreatic cancer or cholangiocarcinoma were screened and enrolled after signing the informed consent forms. In the first stage of the enrolled patients, the 177Lu-EB-FAPI treatment dose was determined using a 3 + 3 dose escalation mode. Patients enrolled in the second phase, divided into pancreatic cancer cohort and cholangiocarcinoma based on pathology, will receive the first phase determined dose of 177Lu-EB-FAPI every 4 weeks, and each patient will receive no more than 4 cycles. The aim of the study is to evaluate the safety and efficacy of the 177Lu-EB-FAPI treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form;
2. Age: 18-75 years old (when signing the informed consent form);
3. Received 68 Ga-FAPI 46 PET imaging positive before treatment;
4. Phase Ia requires patients who have previously failed at least 2 lines of systemic chemotherapy or who the investigator considers unsuitable to receive systemic chemotherapy; Phase Ib Cohort 1, enrollment of patients with hist-or cytologically confirmed metastatic pancreatic cancer; Phase Ib Cohort 2, enrollment of patients with hist-or cytologically confirmed metastatic cholangiocarcinoma;
5. Phase Ia requires at least one evaluable lesion confirmed per RECIST 1.1 criteria; Phase Ib requires at least one measurable lesion confirmed per RECIST 1.1 criteria;
6. ECOG score 0-1, expected survival greater than 3 months;
7. Major organs function well;
8. Patients must have reliable contraception during the study and within 6 months after the study period; negative serum pregnancy / urine pregnancy test within 7 days before study enrollment and must be non-lactating subjects; male subjects should agree to have contraception during the study and within 6 months after the end of the study period.

Exclusion Criteria:

1. Prior treatment before the first dose included chemotherapy and targeted therapy with any associated toxicity (CTCAE v5.0) of> 1 N. A., excluding alopecia;
2. Severe organ failure, such as respiratory failure, uncontrolled thyroid dysfunction including hyperthyroidism and hypothyroidism, or uncorrection of K +, Na +, Ca 2 + electrolyte disorders;
3. Within 5 years, the patient had previous or both other malignant tumors (except for cured skin basal cell carcinoma and cervical carcinoma in situ); had other malignant tumors, but the following two conditions can be enrolled: other malignant tumors treated with single surgery with R0 resection and no recurrence and metastasis; cured cervical carcinoma in situ, skin basal cell carcinoma, nasopharyngeal carcinoma and superficial bladder tumor [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
4. Major surgical treatment with significant traumatic injury within 28 days prior to the first medication;
5. Long-term non-healed wound or fracture; Active bleeding or high risk of bleeding considered by the investigator, such as gastric fundus varices, hemoptysis, etc.;
6. Motor / venous thrombosis events, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, occurred within 6 months before the first medication;
7. Patients with a history of psychiatric substance abuse and unable to quit or with mental disorders;
8. Symptomatic interstitial lung disease, and conditions that may cause drug pulmonary toxicity or associated pneumonia;
9. Patients with any severe and / or uncontrolled disease.
10. Previous history of severe allergy to macromolecular drugs, or allergy to the known component of 177Lu-EB-FAPI injection;
11. Claustrophobic or radiologically phobic patients, or patients with mental disorders or primary affective disorders;
12. According to the discretion of the investigator, subjects with a serious hazard to subject safety or concomitant illness affecting the study or other reasons for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of treatment：hematotoxicity | Up to 2 years.
  Safety evaluation，Complete Blood Count was done continuously during treatment by using CTCAE 5.0 during study
Objective reponse rate (ORR) | Up to 2 years
  The proportion of patients who had tumor evaluated as PR according to RECIST1.1 criteria during phase Ib
Safety of treatment：Hepatotoxicity | Up to 2 years.
  Safety evaluation，liver function lab test was done continuously during treatment and the level of serum ALT, AST, and total bilirubin will be evaluated by using CTCAE 5.0 during study.
Safety of treatment：renal toxicity | Up to 2 years.
  Safety evaluation，renal function lab test was done continuously during treatment and the level of serum creatinine will be evaluated by using CTCAE 5.0 during study.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  The proportion of patients who had tumor evaluated as PR or SD according to RECIST1.1 criteria during phase Ib
Duration of remission （DoR） | Up to 2 years
  The time from the first assessment of the tumor as CR or PR to the first assessment of PD or death from any cause during phase Ib
Progression-free survival （PFS） | Up to 2 years
  The time from enrolled to disease pregression or death from any cause during phase Ib
Overall survival (OS) | Up to 2 years
  The time from enrolled to death from any cause during phase Ib

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No